CLINICAL TRIAL: NCT05423249
Title: Treatment of Non-Anemic Iron Deficiency in Pregnancy: a Double-Blind Randomized Control Trial
Brief Title: Treatment of Non-Anemic Iron Deficiency in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Kimberly Herrera, Clinical Assistant Professor and Associate Maternal Fetal Medicine Fellowship Director, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2022-00121
Record Dates: First submitted 2022-05-19; First posted 2022-06-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Non-anemic Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate; Prenatal Care; Dioctyl Sulfosuccinic Acid; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive oral ferrous sulfate 325mg (containing 65 mg of elemental iron) once daily, an oral prenatal vitamin once daily, oral ascorbic acid 500mg once daily, and oral docusate sodium 100mg twice daily as needed.
  Interventions: Drug: Ferrous sulfate; Drug: Prenatal; Drug: Docusate Sodium; Drug: Ascorbic Acid 500Mg Tab
- Placebo Group (Placebo Comparator): The placebo group will receive a placebo bill, the same oral prenatal vitamin, and oral docusate sodium 100mg twice daily as needed.
  Interventions: Drug: Prenatal; Drug: Docusate Sodium; Drug: Placebo

INTERVENTIONS:
Drug: Ferrous sulfate — Oral ferrous sulfate 325 mg once daily, containing 65 mg of elemental iron to treat non-anemic iron deficiency
  Arms: Treatment Group
Drug: Prenatal — Oral prenatal vitamin once daily for both groups
Drug: Docusate Sodium — Oral docusate sodium 100 mg twice daily as needed, to treat constipation secondary to oral iron supplementation
Drug: Ascorbic Acid 500Mg Tab — Oral ascorbic acid 500 mg daily, to improve absorption of oral iron
  Arms: Treatment Group
Drug: Placebo — Oral placebo pill once daily
  Arms: Placebo Group

SUMMARY:
The objective is to investigate the treatment of non-anemic iron deficiency (NAID) and the impact on development of anemia later in pregnancy. Anemia in the third trimester has been identified as a risk factor for maternal and fetal morbidity that might lead to mortality. Due to the high incidence of NAID in pregnancy, there is an opportunity for early screening and treatment to decrease progression to anemia. The primary aim of this study is to establish if treatment of NAID will result in higher third trimester hemoglobin values and decrease incidence of anemia at term.

DETAILED DESCRIPTION:
All women who fit the inclusion criteria will be approached to be recruited for participation at Stony Brook University Hospital outpatient clinic at less than 20 weeks gestational age. Women who agree to participate in the study will be consented. The study team member will obtain consent from participants and randomize the patient into either the treatment or placebo group based on a 1:1 randomization scheme generated by randomization.com. The study team member will remain blinded, as randomization of subjects will be coordinated by departmental research coordinator, who will not have any interaction with subjects. The treatment group will receive oral ferrous sulfate 325mg (containing 65 mg of elemental iron) daily and a prenatal vitamin, and the placebo group will receive prenatal vitamin and a placebo pill. The prenatal vitamin, which contains iron, will be the same exact formula and will be given to all participants in both control and treatment groups. Only the treatment group will receive the extra iron supplement. The treatment group will also receive vitamin C 500mg daily to assist with iron absorption. Both groups will receive oral docusate sodium (Colace) 100mg twice daily as needed to decrease the risk of constipation.

The randomization will be blinded to the participant, along with the medical provider and study team. Since the Research Pharmacy is able to combine the iron and Vitamin C into one pill, and both groups will receive Colace and prenatal vitamin, the total pill count will not differ from the treatment group and placebo group.

Patients who agree to participate in the study will continue with routine prenatal care and testing, which includes a repeat complete blood count (CBC) in both the second and third trimester, at approximately 24-28 weeks and 34-36 weeks, as is standard of care. In the second and third trimester, a questionnaire will be given to the subject to assess fatigue scores, experience of side effects and severity of side effects. At that time, a study team member will also perform a pill count to assess for compliance.

At time of admission to the hospital for delivery, a repeat ferritin level will be drawn with routine lab work, including a CBC, with no additional risk of blood draw to the patient as this is part of standard of care. The ferritin test will be for research purposes for the study, but will not require an additional blood draw. Clinical anemia will be defined as a hemoglobin level less than or equal to 11 g/dL. While there is no normative data in the literature on ferritin levels in pregnancy, we will define a low ferritin level as <30 mcg/L based on both retrospective pregnancy data and standardized ferritin levels in the non pregnant patient population.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* age 18-55
* less than 20 weeks gestational age
* low ferritin level (<30mcg/L) in the first trimester
* normal hemoglobin level (>11g/dL) in the first trimester

Exclusion Criteria:

* Women with anemia diagnosed in the first trimester (HgB ≤11 g/dL)
* Women with antepartum iron supplementation, except prenatal vitamin, within 3 months
* Women with iron overload or hypersensitivity
* Women with significant vaginal bleeding prior to enrollment
* Women with chronic illness: SLE, hemoglobinopathies, HIV, inflammatory bowel disease, active cancer, prior bariatric surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Delivery admission hemoglobin | From date of randomization until to 42 weeks
  hemoglobin value <11 mg/dL
Third trimester hemoglobin | 28 weeks to 36 weeks
  Incidence of anemia, hemoglobin value <11 mg/dL, in the third trimester

SECONDARY OUTCOMES:
Maternal anemia | Enrollment to 30 days postpartum
  Timing of diagnosis
Incidence of preterm delivery | Enrollment to 30 days postpartum
  Preterm delivery rate
Incidence of maternal hemorrhage | Enrollment to 30 days postpartum
  Postpartum hemorrhage rate
Incidence of treatment of anemia | Enrollment to 30 days postpartum
  Need for IV iron or blood transfusion
Incidence of infection | Enrollment to 30 days postpartum
  infection rate
Maternal hospital stay | Enrollment to 30 days postpartum
  length of hospital stay
Infant weight | Time of birth to 30 days of life
  Birth weight Birth weight, NICU admission, perinatal death
Incidence of neonatal intensive care unit admission | Time of birth to 30 days of life
  Rate of NICU admission Birth weight, NICU admission, perinatal death
Rate of poor perinatal outcome | Time of birth to 30 days of life
  Incidence of perinatal death Birth weight, NICU admission, perinatal death

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University Associates in Obstetrics & Gynecology, Bohemia, New York
  - University Associates in Obstetrics & Gynecology, Commack, New York
  - University Associates in Obstetrics & Gynecology, East Setauket, New York

IPD SHARING:
Plan to Share IPD: No